CLINICAL TRIAL: NCT04048681
Title: Neurological Impacts of Artificial Sweeteners in the Context of Diet Sodas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Olivia Farr, Instructor in Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019P000649
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: artificial sweeteners; diet soda
MeSH Terms: conditions — Obesity | interventions — Coke; Carbonated Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet Soda (Experimental): 12oz can of Diet Coke
  Interventions: Behavioral: diet soda
- Soda (Active Comparator): 12oz can of Coke
  Interventions: Behavioral: Regular soda
- Carbonated Water (Placebo Comparator): 12oz can of carbonated (unflavored) water
  Interventions: Behavioral: Carbonated Water

INTERVENTIONS:
Behavioral: diet soda — 12 oz can of artificially sweetened cola beverage (Diet Coke planned to be used but similar to Diet Pepsi or other Diet Colas)
  Other Names: Diet Coke; Diet Pepsi
  Arms: Diet Soda
Behavioral: Regular soda — 12oz can of regular cola beverage (Coke planned but similar to Pepsi or other regular cola sodas)
  Other Names: Coke; Pepsi
  Arms: Soda
Behavioral: Carbonated Water — 12oz can of carbonated water (sparking water, selzter water) unflavored
  Arms: Carbonated Water

SUMMARY:
This study seeks to determine whether artificial sweeteners in the context of diet soda may alter the brain's response to food cues and thus impact appetite.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are 18-65 years old, with a BMI >30kg/m2.

Exclusion Criteria:

* Unable or unwilling to participate in the study for any reason
* Metal in the body or other safety concerns which makes patient unable to have an MRI
* Pregnant women will be excluded to protect the fetus against potential effects of a non-medically required MRI on fetal development and difficulty of measuring accurate BMI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center MRI Research Facility, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data is HIPAA protected and will not be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross-over trial, and participants were assigned to receive diet soda, regular soda, and carbonated water in a random order.
Groups:
- Diet Soda Then Regular Soda Then Carbonated Water: Participant had first visit with 12oz can of diet soda, 7 days washout, then second visit with 12 oz can of regular soda, 7 days washout, then third visit with 12 oz can of carbonated water.
- Regular Soda Then Carbonated Water Then Diet Soda: Participant had first visit with 12oz can of regular soda, 7 days washout, then second visit with 12 oz can of carbonated water, 7 days washout, then third visit with 12 oz can of diet soda.
- Carbonated Water Then Diet Soda Then Regular Soda: Participant had first visit with 12oz can of carbonated water, 7 days washout, then second visit with 12 oz can of diet soda, 7 days washout, then third visit with 12 oz can of regular soda.
- Regular Soda Then Diet Soda Then Carbonated Water: Participant had first visit with 12oz can of regular soda, 7 days washout, then second visit with 12 oz can of diet soda, 7 days washout, then third visit with 12 oz can of carbonated water.
- Diet Soda Then Carbonated Water Then Regular Soda: Participant had first visit with 12oz can of diet soda, 7 days washout, then second visit with 12 oz can of carbonated water, 7 days washout, then third visit with 12 oz can of regular soda.
Period: Overall Study
Arm/Group | Diet Soda Then Regular Soda Then Carbonated Water | Regular Soda Then Carbonated Water Then Diet Soda | Carbonated Water Then Diet Soda Then Regular Soda | Regular Soda Then Diet Soda Then Carbonated Water | Diet Soda Then Carbonated Water Then Regular Soda
Started | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 0 | 1
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — family emergency | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diet Soda/Regular Soda/ Carbonated Water: The same subjects participated in all three conditions.
Arm/Group | Diet Soda/Regular Soda/ Carbonated Water
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 36.1 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Response to Food Cues in the Insula
Description: Functional magnetic resonance imaging (BOLD signals) while patients view food vs. non-food cues. The effect size z-score represents the magnitude of the activation in that area to food cues vs. non-food cues. The z-score is the estimated response magnitude in that area compared to the overall mean. Negative numbers indicate values lower than the mean and positive numbers indicate values above the mean.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Diet Soda | Soda | Carbonated Water
Number analyzed (Participants) | 5 | 5 | 4
z-score | 0.25 (0.3) | -0.9 (0.3) | -0.01 (0.6)

2. Secondary Outcome: Neurocognitive Testing (Stop Signal Reaction Time)
Description: stop signal reaction time is a measure of inhibitory control, where a shorter stop signal reaction time indicates greater inhibitory control.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: ms
Arm/Group | Diet Soda | Soda | Carbonated Water
Number analyzed (Participants) | 5 | 5 | 4
ms | 162.6 (12.5) | 172.9 (17.4) | 180.2 (19.9)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Diet Soda | Soda | Carbonated Water
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04048681/Prot_SAP_000.pdf